CLINICAL TRIAL: NCT06167746
Title: Improving Care Transitions and Self-care Among Informal Caregivers of Hospitalized Older Adults Through Digital Tools
Brief Title: iCare4Me Transitions
Acronym: iCare4Me T
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: R01AG082892 (NIH); 1R01AG082892-01 (NIH)
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Caregiver Stress
Keywords: Care Transitions; Older Adult; Health Coaching; Virtual; Self-Care; Coping
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Health Information (DHI) (Active Comparator): Digital health information is delivered through a website tailored with care transitions and self-care information for all participants over the 6-month study.
  Interventions: Other: Digital Health Information (DHI)
- Virtual Health Coaching + DHI (Experimental): Study participants in the intervention group will receive 10-session virtual health coaching intervention sessions delivered over 6 months.
  Interventions: Other: Digital Health Information (DHI); Behavioral: Virtual Health Coach for You

INTERVENTIONS:
Other: Digital Health Information (DHI) — Digital health information websites.
Behavioral: Virtual Health Coach for You — Study participants in the intervention group will receive 10-session virtual health coaching intervention session delivered over 6 months with the goal of improving caregiver self-care and coping, decreasing stress, and improving the hospital-to-home experience The 10 sessions are on average 60 minutes and cover the following topics: care transitions, caregiving demand, self-care, and coping.
  Other Names: ViCCY
  Arms: Virtual Health Coaching + DHI

SUMMARY:
The goal of this randomized controlled trial is to examine the effect of a virtual face-to-face health coach intervention to improve self-care among caregivers of hospitalized older adults during care transitions compared to web-based resource information alone to determine the effectiveness of each intervention. The main questions it aims to answer are:

1. compare the efficacy of the virtual health coaching intervention vs. web-based information alone in improving self-care in caregivers of hospitalized community-dwelling older adults with multiple chronic conditions (MCCs) who transition from hospital to home,
2. compare outcomes among Black/African American and White caregivers who receive the intervention vs. digital health information alone, and
3. explore the estimated the cost of the interventions and acute care resource use among patients of caregivers who received virtual intervention vs. digital health information alone.

Participants who enroll will agree to enroll will:

* be randomly assigned to either the health information group or the health coaching intervention plus health information group for six months, and
* be asked to complete a baseline interview, a check-in call at one month post-hospital discharge, and two follow-up interviews at 3- and 6-months after enrollment.

Researchers will compare the two groups of caregivers on the following outcomes: self-care, caregiver self-efficacy (aka confidence), coping, stress, and health status.

ELIGIBILITY:
Inclusion Criteria:

* Informal caregiver providing care at least 8 hours/week to the hospitalized older adult (age 65 or older)
* Reporting poor self-care on screening (Health Self-Care Neglect scale score greater than or equal to 2)
* Willing to use technology (e.g., computer, smartphone, iPad/tablet)
* Able to complete the protocol, e.g., adequate vision and hearing
* English speaking

Exclusion Criteria:

* Cognitive deficits in orientation and/or recall (Six Item Screener score less than 3)
* Participation in another similar support or care transition trial
* Untreated major psychiatric illness (Use of anti-anxiety or anti-depressant medicines is acceptable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Self-Care Inventory | Collected at: enrollment, 3- and 6-months after enrollment
  The Self-Care Inventory (SCI) measures self-care maintenance, monitoring, management, and self-efficacy. Each subscale is standardized on a 0-100 point scale. Higher scores indicate better self-care.
Health Self-Care Neglect | Collected at: enrollment, 3- and 6-months after enrollment
  This a binary that scale captures the level of self-care neglect, with higher scores indicating greater neglect.

SECONDARY OUTCOMES:
Perceived Stress Scale | Collected at: enrollment, 3- and 6-months after enrollment
  The perceived stress scale has 10 items rated on a 5-point scale rating perceptions of stress.
Brief COPE | Collected at: enrollment, 3- and 6-months after enrollment
  This tool is designed to assess the varying coping strategies used by individuals in response to stress.
Caregiver Self-Care Self-Efficacy Scale | Collected at: enrollment, 3- and 6-months after enrollment
  This scale measures caregiving self-efficacy in multiple areas. Each item is measured on a scale of 1-5 with 5 indicating they are the most confident in that area.
Preparedness for Caregiving Scale | Collected at: enrollment, 3- and 6-months after enrollment
  This scale measures how prepared caregivers feel to provide support for their loved ones in multiple areas. Each item is measured on a scale of 0-4 with 4 indicating they are the most prepared in that area.
Quality of the relationship | Collected at: enrollment, 3- and 6-months after enrollment
  This scale measures giving and receiving support in multiple areas. Each item is measured on a scale of 0-4 with 4 indicating they are the most positive in that area.
RAND Medical Outcomes Study Short Form (SF-36) | Collected at: enrollment, 3- and 6-months after enrollment
  This scale that uses multiple measures to determine overall mental and physical health. Higher scores indicate better mental and physical health.

OTHER OUTCOMES:
Experience with Care | Collected at 1 month post index-hospital discharge
  This 10-item tool evaluates the experience with care post-hospital discharge. Each item is measured on a scale of 1-4 with 4 indicating they strongly agree with each statement.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Hirschman, Ph.D., Principal Investigator — University of Pennsylvia
Locations (3):
- United States (3):
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Individual participant self-report data collected during the trial that underlie the results of the primary outcome will be shared after de-identification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available as soon as possible but no later than within one year of the completion of the funded project period for the parent award or upon acceptance of the data for publication, whichever is earlier. Data will be preserved for at least five years following the end of the grant period.
Access Criteria: Individual-level data will be shared with controlled access as allowed by informed consent agreements approved by the University of Pennsylvania Institutional Review Board (IRB). Data sharing and confidentiality agreements as established by the university or future data repository will be required.